CLINICAL TRIAL: NCT00002177
Title: A Pilot Open Label Trial of HIV Therapy With d4T (Stavudine), ddI (Didanosine), Nelfinavir and Hydroxyurea in Subjects With Recent HIV Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 244D; AI455-063
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2011-04

CONDITIONS: HIV Infections
Keywords: Pilot Projects; HIV-1; Didanosine; Drug Therapy, Combination; Stavudine; Hydroxyurea; RNA, Viral; Nelfinavir; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Hydroxyurea; Nelfinavir; Stavudine; Didanosine

INTERVENTIONS:
Drug: Hydroxyurea
Drug: Nelfinavir mesylate
Drug: Stavudine
Drug: Didanosine

SUMMARY:
To assess the magnitude and duration of the antiviral activity in plasma and the incidence and time to total suppression of detectable HIV RNA in plasma. To assess the long-term safety and tolerability of this combination therapy and the magnitude and duration of the effect of these drugs over CD4 cell counts.

ELIGIBILITY:
Inclusion Criteria

Patients must have the following symptoms and conditions:

* Treatment naive.
* Recent HIV infection.
* Baseline laboratory values within acceptable ranges.
* Written, informed consent from parent or legal guardian for patients < 18 years old.
* Available for follow-up for at least 96 weeks.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions and symptoms are excluded:

* Documentation of other cause for previously mentioned clinical conditions.
* Intractable diarrhea.
* Signs and symptoms of bilateral peripheral neuropathy >= Grade 2.
* Inability to tolerate oral medication.
* Hemophilia, other bleeding disorder, or no accessible tonsillar or lymph node tissue.

Patients with the following prior conditions are excluded:

History of acute or chronic pancreatitis. 1. Use of potent neurotoxic drugs is not permitted.

* No other anti-HIV therapy allowed.
* Nelfinavir should not be administered concurrently with rifampin or rifabutin, terfenadine (Seldane), astemizole (Hismanal), cisapride (Propulsid), triazolam (Halcion), and midazolam (Versed).

  1. Any prior antiretroviral therapy.
* Prior vaccination with a candidate HIV therapeutic vaccine.
* Previous therapy with agents with significant systemic myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic or cytotoxic potential within 3 months of study start or the expected need for such therapy at the time of enrollment.
* Previous therapy with rifampin or rifabutin, terfenadine (Seldane), astemizole (Hismanal), cisapride (Propulsid), triazolam (Halcion), and midazolam (Versed) within 14 days prior to study entry or at any time while on study.

Active alcohol or substance abuse.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-05; Primary Completion 2000-03 (Actual); Study Completion 2000-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of California at San Francisco Gen Hosp, San Francisco, California, United States